CLINICAL TRIAL: NCT00942097
Title: Homeopathic Treatment in Pregnant Women With Overweight and Mental Disorder: a Double Blinded Controlled Clinical Trial
Brief Title: Homeopathic Medication and Nutritional Oriented Diet to Treat Overweight Pregnant Women With Mental Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Edgard Costa de Vilhena (Other)
Collaborators: Amparo Maternal Maternidade Social (Other)
Responsible Party: Sponsor-Investigator, Edgard Costa de Vilhena, MD, student PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HAM-01082009; Homeopathy (Other: 6904562)
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Overweight; Pregnancy; Mental Disorder
Keywords: Homeopathy; overweight; obesity; mental disorder; pregnancy; Overweight pregnant women with suspicious mental disorder
MeSH Terms: conditions — Overweight; Mental Disorders; Obesity | interventions — Selenoprotein P; Phosphorus, Dietary; Sulfur; Phosphorus; Homeopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional plus Placebo (homeopathy) (Placebo Comparator): Nutritional oriented diet for pregnancy period add homeopathic preparation from inert substance.
  Interventions: Drug: Sulph, Puls, Lyc, Lack t, Con, Sep, Nux v, Calc c, Phos; Drug: Homeopathy and Nutritional oriented diet
- Nutr and Homeop Sulph Puls Lyc Lackt Con Sep Nuxv Calcc Phos (Active Comparator): Nutrition oriented diet for pregnancy period add active homeopathic medication (Sulph, Puls, Lyc, Lack t, Con, Sep, Nux v, Calc c, Phos)
  Interventions: Drug: Sulph, Puls, Lyc, Lack t, Con, Sep, Nux v, Calc c, Phos; Drug: Homeopathy and Nutritional oriented diet

INTERVENTIONS:
Drug: Sulph, Puls, Lyc, Lack t, Con, Sep, Nux v, Calc c, Phos — CH 12 preparation, 6 drops, twice a day, 4 days per week, until the end of pregnancy. One medication per appointment.
  Other Names: Sulphur; Puls; Lyc; Lack-t; Conium-m; Nux-v; Calc-c; Sep; Phosphorus
Drug: Homeopathy and Nutritional oriented diet — Homeopathy 6 drops twice a day 4 days per week, active and placebo and Balanced nutritional oriented diet for both groups.

SUMMARY:
The purpose of this study is to evaluate the efficacy of homeopathic treatment in pregnant women with overweight and class I obesity with suspicion of a mental disorder.

DETAILED DESCRIPTION:
The weight gain during pregnancy has been reported as an important factor of being overweight after delivery and comorbidities. There are a lot of restrictions to treat pregnant women due to fetus development. Homeopathy presents itself as an integrative medicine that could treat with less collateral effects improving general health. The investigators are going to test the effects of homeopathy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with less than 28 weeks,
* BMI from 26 to 35 Kg/ m2,
* SRQ-20 positive.

Exclusion Criteria:

* Diabetes
* Cardiopathies
* Hypertension
* Nephropathies
* Psychiatric treatment
* Drug users
* Pulmonary Chronic Disease
* Suicidal ideas
* No eating (appetites)
* Problems of BMI measurements (disabled people)
* Concomitant homeopathic treatment
* People who are looking for just 1 medical appointment

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Weight | 9 months

SECONDARY OUTCOMES:
Comorbidities | 9 months
Newborn weight | 9 months
Pregnancy period | 9 months
Collateral effects | 9 months
Self perception health | 9 months
Apgar score | 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Edgard C Vilhena, MD, Principal Investigator — Medicine School - University of São Paulo
Locations (1):
- Amparo Maternal Maternidade Social, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Keppel KG, Taffel SM. Pregnancy-related weight gain and retention: implications of the 1990 Institute of Medicine guidelines. Am J Public Health. 1993 Aug;83(8):1100-3. doi: 10.2105/ajph.83.8.1100. PMID 8342716
- [Background] Horton R. The neglected epidemic of chronic disease. Lancet. 2005 Oct 29-Nov 4;366(9496):1514. doi: 10.1016/S0140-6736(05)67454-5. No abstract available. PMID 16257331
- [Background] Strong K, Mathers C, Leeder S, Beaglehole R. Preventing chronic diseases: how many lives can we save? Lancet. 2005 Oct 29-Nov 4;366(9496):1578-82. doi: 10.1016/S0140-6736(05)67341-2. PMID 16257345
- [Background] Fuster V, Voute J. MDGs: chronic diseases are not on the agenda. Lancet. 2005 Oct 29-Nov 4;366(9496):1512-4. doi: 10.1016/S0140-6736(05)67610-6. No abstract available. PMID 16257330
- [Background] Monteiro CA, Conde WL, Popkin BM. Is obesity replacing or adding to undernutrition? Evidence from different social classes in Brazil. Public Health Nutr. 2002 Feb;5(1A):105-12. doi: 10.1079/PHN2001281. PMID 12027272
- [Background] Yang D, Fontaine KR, Wang C, Allison DB. Weight loss causes increased mortality: cons. Obes Rev. 2003 Feb;4(1):9-16. doi: 10.1046/j.1467-789x.2003.00092.x. PMID 12608523
- [Background] Hubert HB, Feinleib M, McNamara PM, Castelli WP. Obesity as an independent risk factor for cardiovascular disease: a 26-year follow-up of participants in the Framingham Heart Study. Circulation. 1983 May;67(5):968-77. doi: 10.1161/01.cir.67.5.968. PMID 6219830
- [Background] Frankel PH. Obesity and cancer. N Engl J Med. 2003 Jul 31;349(5):502-4; author reply 502-4. No abstract available. PMID 12892102
- [Background] Allison DB, Saunders SE. Obesity in North America. An overview. Med Clin North Am. 2000 Mar;84(2):305-32, v. doi: 10.1016/s0025-7125(05)70223-6. PMID 10793644
- [Background] Allison DB, Fontaine KR, Manson JE, Stevens J, VanItallie TB. Annual deaths attributable to obesity in the United States. JAMA. 1999 Oct 27;282(16):1530-8. doi: 10.1001/jama.282.16.1530. PMID 10546692
- [Background] Harris T, Cook EF, Garrison R, Higgins M, Kannel W, Goldman L. Body mass index and mortality among nonsmoking older persons. The Framingham Heart Study. JAMA. 1988 Mar 11;259(10):1520-4. PMID 3339789
- [Background] Chu SY, Callaghan WM, Kim SY, Schmid CH, Lau J, England LJ, Dietz PM. Maternal obesity and risk of gestational diabetes mellitus. Diabetes Care. 2007 Aug;30(8):2070-6. doi: 10.2337/dc06-2559a. Epub 2007 Apr 6. PMID 17416786
- [Background] Ohlin A, Rossner S. Maternal body weight development after pregnancy. Int J Obes. 1990 Feb;14(2):159-73. PMID 2341224
- [Background] Greene GW, Smiciklas-Wright H, Scholl TO, Karp RJ. Postpartum weight change: how much of the weight gained in pregnancy will be lost after delivery? Obstet Gynecol. 1988 May;71(5):701-7. PMID 3357658
- [Background] Linne Y, Barkeling B, Rossner S. Long-term weight development after pregnancy. Obes Rev. 2002 May;3(2):75-83. doi: 10.1046/j.1467-789x.2002.00061.x. PMID 12120423
- [Background] Gore SA, Brown DM, West DS. The role of postpartum weight retention in obesity among women: a review of the evidence. Ann Behav Med. 2003 Oct;26(2):149-59. doi: 10.1207/S15324796ABM2602_07. PMID 14534032
- [Background] Lederman SA. Pregnancy weight gain and postpartum loss: avoiding obesity while optimizing the growth and development of the fetus. J Am Med Womens Assoc (1972). 2001 Spring;56(2):53-8. PMID 11326797
- [Background] Boardley DJ, Sargent RG, Coker AL, Hussey JR, Sharpe PA. The relationship between diet, activity, and other factors, and postpartum weight change by race. Obstet Gynecol. 1995 Nov;86(5):834-8. doi: 10.1016/0029-7844(95)00283-W. PMID 7566859
- [Background] Parker JD, Abrams B. Differences in postpartum weight retention between black and white mothers. Obstet Gynecol. 1993 May;81(5 ( Pt 1)):768-74. PMID 8469470
- [Background] Potter S, Hannum S, McFarlin B, Essex-Sorlie D, Campbell E, Trupin S. Does infant feeding method influence maternal postpartum weight loss? J Am Diet Assoc. 1991 Apr;91(4):441-6. PMID 2016492
- [Background] Scholl TO, Hediger ML, Schall JI, Ances IG, Smith WK. Gestational weight gain, pregnancy outcome, and postpartum weight retention. Obstet Gynecol. 1995 Sep;86(3):423-7. doi: 10.1016/0029-7844(95)00190-3. PMID 7651655
- [Background] Bradley PJ. Conditions recalled to have been associated with weight gain in adulthood. Appetite. 1985 Sep;6(3):235-41. PMID 4073883
- [Background] Hill JO, Peters JC. Environmental contributions to the obesity epidemic. Science. 1998 May 29;280(5368):1371-4. doi: 10.1126/science.280.5368.1371. PMID 9603719
- [Background] Maddi SR, Khoshaba DM, Persico M, Bleecker F, VanArsdall G. Psychosocial correlates of psychopathology in a national sample of the morbidly obese. Obes Surg. 1997 Oct;7(5):397-404. doi: 10.1381/096089297765555377. PMID 9730493
- [Background] Lundberg U, Frankenhaeuser M. Pituitary-adrenal and sympathetic-adrenal correlates of distress and effort. J Psychosom Res. 1980;24(3-4):125-30. doi: 10.1016/0022-3999(80)90033-1. No abstract available. PMID 7441580
- [Background] Pop-Jordanova N. Psychological characteristics and biofeedback mitigation in preadolescents with eating disorders. Pediatr Int. 2000 Feb;42(1):76-81. doi: 10.1046/j.1442-200x.2000.01176.x. PMID 10703241
- [Background] Coggon D, Martyn C, Palmer KT, Evanoff B. Assessing case definitions in the absence of a diagnostic gold standard. Int J Epidemiol. 2005 Aug;34(4):949-52. doi: 10.1093/ije/dyi012. PMID 16076861
- [Background] Botega NJ, Bio MR, Zomignani MA, Garcia C Jr, Pereira WA. [Mood disorders among inpatients in ambulatory and validation of the anxiety and depression scale HAD]. Rev Saude Publica. 1995 Oct;29(5):355-63. doi: 10.1590/s0034-89101995000500004. Portuguese. PMID 8731275
- [Background] Kessler RC, Molnar BE, Feurer ID, Appelbaum M. Patterns and mental health predictors of domestic violence in the United States: results from the National Comorbidity Survey. Int J Law Psychiatry. 2001 Jul-Oct;24(4-5):487-508. doi: 10.1016/s0160-2527(01)00080-2. No abstract available. PMID 11521422
- [Background] Kendler KS, Neale MC, Kessler RC, Heath AC, Eaves LJ. Major depression and generalized anxiety disorder. Same genes, (partly) different environments? Arch Gen Psychiatry. 1992 Sep;49(9):716-22. doi: 10.1001/archpsyc.1992.01820090044008. PMID 1514877
- [Background] Pine DS, Cohen P, Gurley D, Brook J, Ma Y. The risk for early-adulthood anxiety and depressive disorders in adolescents with anxiety and depressive disorders. Arch Gen Psychiatry. 1998 Jan;55(1):56-64. doi: 10.1001/archpsyc.55.1.56. PMID 9435761
- [Background] Wittchen HU, Stein MB, Kessler RC. Social fears and social phobia in a community sample of adolescents and young adults: prevalence, risk factors and co-morbidity. Psychol Med. 1999 Mar;29(2):309-23. doi: 10.1017/s0033291798008174. PMID 10218923
- [Background] McCarter-Spaulding DE. Medications in pregnancy and lactation. MCN Am J Matern Child Nurs. 2005 Jan-Feb;30(1):10-7; quiz 18-9. PMID 15622140
- [Background] Fisher P, Ward A. Complementary medicine in Europe. BMJ. 1994 Jul 9;309(6947):107-11. doi: 10.1136/bmj.309.6947.107. PMID 8038643
- [Background] Endler PC, Pongratz W, Smith CW, Schulte J. Non-molecular information transfer from thyroxine to frogs with regard to homeopathic toxicology. Vet Hum Toxicol. 1995 Jun;37(3):259-60. No abstract available. PMID 7571362
- [Background] Dugoua JJ, Mills E, Perri D, Koren G. Safety and efficacy of St. John's wort (hypericum) during pregnancy and lactation. Can J Clin Pharmacol. 2006 Fall;13(3):e268-76. Epub 2006 Nov 3. PMID 17085775
- [Background] McKenna L, McIntyre M. What over-the-counter preparations are pregnant women taking? A literature review. J Adv Nurs. 2006 Dec;56(6):636-45. doi: 10.1111/j.1365-2648.2006.04037.x. PMID 17118042
- [Background] Field T. Pregnancy and labor alternative therapy research. Altern Ther Health Med. 2008 Sep-Oct;14(5):28-34. PMID 18780582
- [Background] Dayan J, Yoshida K. [Psychological and pharmacological treatments of mood and anxiety disorders during pregnancy and postpartum. Review and synthesis]. J Gynecol Obstet Biol Reprod (Paris). 2007 Oct;36(6):530-48. doi: 10.1016/j.jgyn.2007.06.004. Epub 2007 Jul 5. French. PMID 17616265
- [Background] Charlton RA, Cunnington MC, de Vries CS, Weil JG. Data resources for investigating drug exposure during pregnancy and associated outcomes: the General Practice Research Database (GPRD) as an alternative to pregnancy registries. Drug Saf. 2008;31(1):39-51. doi: 10.2165/00002018-200831010-00004. PMID 18095745
- [Background] Kyle PM. Drugs and the fetus. Curr Opin Obstet Gynecol. 2006 Apr;18(2):93-9. doi: 10.1097/01.gco.0000192974.61729.4c. PMID 16601467
- [Background] Guelinckx I, Devlieger R, Beckers K, Vansant G. Maternal obesity: pregnancy complications, gestational weight gain and nutrition. Obes Rev. 2008 Mar;9(2):140-50. doi: 10.1111/j.1467-789X.2007.00464.x. Epub 2008 Jan 21. PMID 18221480
- [Background] Polley BA, Wing RR, Sims CJ. Randomized controlled trial to prevent excessive weight gain in pregnant women. Int J Obes Relat Metab Disord. 2002 Nov;26(11):1494-502. doi: 10.1038/sj.ijo.0802130. PMID 12439652
- [Background] Pearlstein T. Perinatal depression: treatment options and dilemmas. J Psychiatry Neurosci. 2008 Jul;33(4):302-18. PMID 18592032
- [Background] Bonari L, Pinto N, Ahn E, Einarson A, Steiner M, Koren G. Perinatal risks of untreated depression during pregnancy. Can J Psychiatry. 2004 Nov;49(11):726-35. doi: 10.1177/070674370404901103. PMID 15633850
- [Background] Epstein LH, Wing RR, Penner BC, Kress MJ. Effect of diet and controlled exercise on weight loss in obese children. J Pediatr. 1985 Sep;107(3):358-61. doi: 10.1016/s0022-3476(85)80506-0. PMID 4032130
- [Background] Harding TW, de Arango MV, Baltazar J, Climent CE, Ibrahim HH, Ladrido-Ignacio L, Murthy RS, Wig NN. Mental disorders in primary health care: a study of their frequency and diagnosis in four developing countries. Psychol Med. 1980 May;10(2):231-41. doi: 10.1017/s0033291700043993. PMID 7384326
- [Background] Mari JJ, Williams P. A comparison of the validity of two psychiatric screening questionnaires (GHQ-12 and SRQ-20) in Brazil, using Relative Operating Characteristic (ROC) analysis. Psychol Med. 1985 Aug;15(3):651-9. doi: 10.1017/s0033291700031500. PMID 4048323
- [Background] Mari JJ, Williams P. A validity study of a psychiatric screening questionnaire (SRQ-20) in primary care in the city of Sao Paulo. Br J Psychiatry. 1986 Jan;148:23-6. doi: 10.1192/bjp.148.1.23. PMID 3955316
- [Background] Milgrom LR. Vitalism, complexity and the concept of spin. Homeopathy. 2002 Jan;91(1):26-31. doi: 10.1054/homp.2001.0013. PMID 12371447
- [Background] Milgrom LR. Patient-practitioner-remedy (PPR) entanglement. Part 3. Refining the quantum metaphor for homeopathy. Homeopathy. 2003 Jul;92(3):152-60. doi: 10.1016/s1475-4916(03)00038-9. PMID 12884898
- [Background] Teixeira MZ. Homeopathic use of modern medicines: utilisation of the curative rebound effect. Med Hypotheses. 2003 Feb;60(2):276-83. doi: 10.1016/s0306-9877(02)00386-9. PMID 12606247
- [Background] Weingartner O. What is the therapeutically active ingredient of homeopathic potencies? Homeopathy. 2003 Jul;92(3):145-51. doi: 10.1016/s1475-4916(03)00037-7. PMID 12884897
- [Background] Linde K, Clausius N, Ramirez G, Melchart D, Eitel F, Hedges LV, Jonas WB. Are the clinical effects of homeopathy placebo effects? A meta-analysis of placebo-controlled trials. Lancet. 1997 Sep 20;350(9081):834-43. doi: 10.1016/s0140-6736(97)02293-9. PMID 9310601
- [Background] Shang A, Huwiler-Muntener K, Nartey L, Juni P, Dorig S, Sterne JA, Pewsner D, Egger M. Are the clinical effects of homoeopathy placebo effects? Comparative study of placebo-controlled trials of homoeopathy and allopathy. Lancet. 2005 Aug 27-Sep 2;366(9487):726-32. doi: 10.1016/S0140-6736(05)67177-2. PMID 16125589
- [Background] Oberbaum M, Singer SR, Frass M. Homeopathic research after the Lancet meta analysis--a moment for introspection. Complement Ther Med. 2005 Dec;13(4):303-5. doi: 10.1016/j.ctim.2005.10.006. Epub 2005 Nov 17. No abstract available. PMID 16338202
- [Background] Mathie RT. The research evidence base for homeopathy: a fresh assessment of the literature. Homeopathy. 2003 Apr;92(2):84-91. doi: 10.1016/s1475-4916(03)00006-7. PMID 12725250
- [Background] Jonas WB, Kaptchuk TJ, Linde K. A critical overview of homeopathy. Ann Intern Med. 2003 Mar 4;138(5):393-9. doi: 10.7326/0003-4819-138-5-200303040-00009. PMID 12614092
- [Background] White A, Slade P, Hunt C, Hart A, Ernst E. Individualised homeopathy as an adjunct in the treatment of childhood asthma: a randomised placebo controlled trial. Thorax. 2003 Apr;58(4):317-21. doi: 10.1136/thorax.58.4.317. PMID 12668794
- [Background] Jacobs J, Springer DA, Crothers D. Homeopathic treatment of acute otitis media in children: a preliminary randomized placebo-controlled trial. Pediatr Infect Dis J. 2001 Feb;20(2):177-83. doi: 10.1097/00006454-200102000-00012. PMID 11224838
- [Background] Frei H, Thurneysen A. Homeopathy in acute otitis media in children: treatment effect or spontaneous resolution? Br Homeopath J. 2001 Oct;90(4):180-2. doi: 10.1054/homp.1999.0505. PMID 11680801
- [Background] Taylor MA, Reilly D, Llewellyn-Jones RH, McSharry C, Aitchison TC. Randomised controlled trial of homoeopathy versus placebo in perennial allergic rhinitis with overview of four trial series. BMJ. 2000 Aug 19-26;321(7259):471-6. doi: 10.1136/bmj.321.7259.471. PMID 10948025
- [Background] Jacobs J, Jonas WB, Jimenez-Perez M, Crothers D. Homeopathy for childhood diarrhea: combined results and metaanalysis from three randomized, controlled clinical trials. Pediatr Infect Dis J. 2003 Mar;22(3):229-34. doi: 10.1097/01.inf.0000055096.25724.48. PMID 12634583
- [Background] Frass M, Linkesch M, Banyai S, Resch G, Dielacher C, Lobl T, Endler C, Haidvogl M, Muchitsch I, Schuster E. Adjunctive homeopathic treatment in patients with severe sepsis: a randomized, double-blind, placebo-controlled trial in an intensive care unit. Homeopathy. 2005 Apr;94(2):75-80. doi: 10.1016/j.homp.2005.01.002. PMID 15892486
- [Background] Olson CM. Achieving a healthy weight gain during pregnancy. Annu Rev Nutr. 2008;28:411-23. doi: 10.1146/annurev.nutr.28.061807.155322. PMID 18422452
- [Background] Kiel DW, Dodson EA, Artal R, Boehmer TK, Leet TL. Gestational weight gain and pregnancy outcomes in obese women: how much is enough? Obstet Gynecol. 2007 Oct;110(4):752-8. doi: 10.1097/01.AOG.0000278819.17190.87. PMID 17906005
- [Background] Idler EL, Benyamini Y. Self-rated health and mortality: a review of twenty-seven community studies. J Health Soc Behav. 1997 Mar;38(1):21-37. PMID 9097506
- See also: Groupe International de Recherche sur l'infinitesimal — http://giriweb.com
- See also: Homeopathé International — http://www.homeoint.org
- See also: Morpho logica Homeopatica Ruby — http://www.morphologica.com